CLINICAL TRIAL: NCT02266134
Title: Standardized Versus Tailored Implementation of Measurement Based Care for Depression
Acronym: iMBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Lewis, Associate Investigator, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1R01MH103310-01A1 (NIH)
Record Dates: First submitted 2014-10-12; First posted 2014-10-16 (Estimated); Results first posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Depression
Keywords: implementation; measurement based care; standardized; tailored
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standardized Implementation, Patients (Experimental): Sites in standardized condition arm will receive the standard implementation of measurement-based care intervention (PHQ-9).
  Interventions: Behavioral: Standard Implementation of Measurement Based Care
- Tailored Implementation, Patients (Experimental): Sites in the tailored condition arm will receive the tailored implementation of measurement-based care intervention (PHQ-9).
  Interventions: Behavioral: Tailored Implementation of Measurement Based Care
- Standardized Implementation, Therapists (Experimental): Sites randomized to the standardized condition will be expected to use the measurement-based care intervention (PHQ-9) prior to each session with a depressed client and they will work as a team to maximize fidelity.
  Interventions: Behavioral: Standard Implementation of Measurement Based Care
- Tailored Implementation, Therapists (Experimental): Sites randomized to the tailored condition will develop a site-specific protocol for use of the measurement-based care intervention (PHQ-9), and they will work as a team to maximize the fit of measurement-based care to this clinic.
  Interventions: Behavioral: Tailored Implementation of Measurement Based Care

INTERVENTIONS:
Behavioral: Tailored Implementation of Measurement Based Care — Measurement-based care in this study is the practice of basing psychotherapeutic services on the results of the Patient Health Questionnaire; the implementation of measurement-based care will be tailored based on clinic specific barriers and facilitators.
  Arms: Tailored Implementation, Patients; Tailored Implementation, Therapists
Behavioral: Standard Implementation of Measurement Based Care — Measurement-based care in this study is the practice of basing psychotherapeutic services on the results of the Patient Health Questionnaire (PHQ-9); the implementation of measurement-based care will be standardized such that clinicians will be encouraged to administer the PHQ-9 to depressed clients before each session.
  Arms: Standardized Implementation, Patients; Standardized Implementation, Therapists

SUMMARY:
Depression remains among the nation's top 10 chronic illnesses, costing over $80 billion annually; however, Measurement Based Care (MBC) is a relatively simple evidence-based intervention framework that has been shown to improve outcomes for depressed clients by identifying those who are not making progress and reducing the likelihood that clients will deteriorate in treatment. Despite the demonstrated effectiveness of MBC, the majority of community mental health counselors do not regularly assess target problem symptoms to guide their work. This study will test a standardized versus a tailored approach to implementing MBC that will include the integration of symptom monitoring capacities into the electronic health record system of one of the nation's largest not-for-profit providers of behavioral health services.

DETAILED DESCRIPTION:
Depression remains among the nation's top 10 chronic illnesses, costing over $80 billion annually. Depression has been called the "Common Cold" of mental illness, but one with serious risk of morbidity and mortality. There are now many evidence-based practices for the treatment of depression, but unfortunately these practices remain largely unavailable to clients receiving services in community mental health centers. Measurement Based Care (MBC) is a relatively simple evidence-based intervention framework. MBC, by definition, is the practice of using symptom measurement to inform mental health care. Physicians who routinely measure the patient's blood pressure when the treatment target is high blood pressure demonstrate the medical corollary of MBC. When MBC is used in the treatment of depressed adults, it has been shown to improve outcomes by identifying clients who are not making progress and reducing the likelihood that clients will deteriorate in treatment. However, despite the demonstrated effectiveness of MBC, the majority of community mental health counselors (i.e., clinicians) do not regularly assess target problem symptoms to guide their work over the course of treatment. To our knowledge, no studies to date have focused on the process of implementing MBC in community mental health settings. The long-term goal of this research project is to provide generalizable and practical recommendations about implementation approaches that promote MBC use and fidelity in community mental health centers. Specifically, this study will test a standardized versus a tailored approach to implementing MBC in one of the nation's largest not-for-profit providers of behavioral health services. Although touted as superior, tailored implementations have rarely been compared to standardized approaches. Moreover, recent research has demonstrated an apparent need to adapt evidence-based practices to fit the specific context in which they are being implemented, particularly if they are to be sustained. This proposal reflects a movement in the field of implementation science in which planned adaptations are being tested and compared to standardized versions. The proposed research is a three-phase, mixed methods (quantitative/qualitative) study to investigate the effect of these two different approaches to MBC implementation on both clinician-level (e.g., MBC fidelity) and client-level (depression symptom change) outcomes. We will focus on contextual factors (e.g., attitudes, resources, process, etc.) that may influence the implementation process with the goal of identifying a generalizable and practical way of bringing MBC to community mental health centers treating depressed adults.

ELIGIBILITY:
To be included, Patients must:

1. be age 18 or above at time of enrollment;
2. have depression as one of their primary treatment foci based on diagnosis made by clinicians using usual care interview methods to reflect major depressive disorder, dysthymic disorder, depressive disorder NOS, adjustment disorder with depressed mood;
3. have significant depressive symptom severity (PHQ-9 total score > 9);
4. receive individual psychotherapy;
5. be fluent in English; and
6. receive therapy from an enrolled study clinician during the proposed funding period

Patients will be excluded if they have an inability to sign the consent form (due to lack of competence or inability to read).

Therapist Inclusion Criteria -- Therapists must:

1. be a practicing clinician at Centerstone; and
2. see at least one adult (18+) patient

Therapist Exclusion Criteria: N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cara C Lewis, PhD, Principal Investigator — Indiana University
Locations (6):
- United States (6):
  - Centerstone Connersville, Connersville, Indiana
  - Centerstone Martinsville, Martinsville, Indiana
  - Centerstone Columbia, Columbia, Tennessee
  - Centerstone Dede Wallace Campus, Nashville, Tennessee
  - Centerstone Frank Luton Center, Nashville, Tennessee
  - Centerstone Tullahoma, Tullahoma, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Snider MDH, Boyd MR, Walker MR, Powell BJ, Lewis CC. Using audit and feedback to guide tailored implementations of measurement-based care in community mental health: a multiple case study. Implement Sci Commun. 2023 Aug 14;4(1):94. doi: 10.1186/s43058-023-00474-8. PMID 37580815
- [Derived] Lewis CC, Boyd MR, Marti CN, Albright K. Mediators of measurement-based care implementation in community mental health settings: results from a mixed-methods evaluation. Implement Sci. 2022 Oct 21;17(1):71. doi: 10.1186/s13012-022-01244-1. PMID 36271404
- [Derived] Albright K, Navarro EI, Jarad I, Boyd MR, Powell BJ, Lewis CC. Communication strategies to facilitate the implementation of new clinical practices: a qualitative study of community mental health therapists. Transl Behav Med. 2022 Feb 16;12(2):324-334. doi: 10.1093/tbm/ibab139. PMID 34791490
- [Derived] Lewis CC, Scott K, Marti CN, Marriott BR, Kroenke K, Putz JW, Mendel P, Rutkowski D. Implementing measurement-based care (iMBC) for depression in community mental health: a dynamic cluster randomized trial study protocol. Implement Sci. 2015 Sep 7;10:127. doi: 10.1186/s13012-015-0313-2. PMID 26345270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 community-based behavioral health clinics were randomized into four groups: (1) Sites 1-2; (2) Sites 3-6; (3) Sites 7-10; and (4) Sites 11-12.
  Therapist recruitment was in-person or via email from June 3, 2015-October 18, 2016.
  Patient recruitment was staggered such that each site began recruitment approximately five months apart. Recruitment start dates: (1) Sites 1-2: August 13, 2015; Sites 3-6: December 7, 2015; Sites 7-10: May 20, 2016; and Sites 11-12: December 2, 2016.
Pre-assignment Details: Of the 2459 patients assessed for eligibility, 228 met inclusion criteria and were enrolled during the study's active implementation window (0-5 months).
  Of the 525 therapists assessed for eligibility, 154 met inclusion criteria and consented during the study's active implementation window (0-5 months).
Units Other Than Participants: Health Clinics
Groups:
- Standardized Implementation, Patients: Sites in the standardized condition arm will receive the standard implementation of measurement-based care intervention (PHQ-9).
- Tailored Implementation, Patients: Sites randomized to the tailored condition will develop a site-specific protocol for use of the Patient Health Questionnaire and they will work as a team to maximize the fit of measurement based care to this clinic.
- Standardized Implementation, Therapists: Sites randomized to the standardized condition will be expected to use the Patient Health Questionnaire prior to each session with a depressed client, and they will work as a team to maximize fidelity.
- Tailored Condition, Therapists: Sites in the tailored condition will develop a site-specific protocol for use of the Patient Health Questionnaire and they will work as a team to maximize the fit of measurement-based care to tailored clinic.
Period: Clinics #1-2: Beginning Aug 2015
Arm/Group | Standardized Implementation, Patients | Tailored Implementation, Patients | Standardized Implementation, Therapists | Tailored Condition, Therapists
Started | 9; 1 Health Clinics | 11; 1 Health Clinics | 14; 1 Health Clinics | 14; 1 Health Clinics
Completed (For patients, completion of the study refers to patients who completed both a baseline PHQ-9 and a 12-week PHQ-9. For therapists, completion of the study refers to therapists who completed a baseline assessment and contributed to PHQ-9 fidelity data.) | 3; 1 Health Clinics | 8; 1 Health Clinics | 14; 1 Health Clinics | 14; 1 Health Clinics
Not Completed | 6; 0 Health Clinics | 3; 0 Health Clinics | 0; 0 Health Clinics | 0; 0 Health Clinics
Not completed — Lost to Follow-up | 6 | 3 | 0 | 0
Period: Clinics #3-6: Beginning Dec 2015
Arm/Group | Standardized Implementation, Patients | Tailored Implementation, Patients | Standardized Implementation, Therapists | Tailored Condition, Therapists
Started | 47; 2 Health Clinics | 24; 2 Health Clinics | 14; 2 Health Clinics | 17; 2 Health Clinics
Completed | 39; 2 Health Clinics | 22; 2 Health Clinics | 14; 2 Health Clinics | 17; 2 Health Clinics
Not Completed | 8; 0 Health Clinics | 2; 0 Health Clinics | 0; 0 Health Clinics | 0; 0 Health Clinics
Not completed — Lost to Follow-up | 8 | 2 | 0 | 0
Period: Clinics #7-10: Beginning May 2016
Arm/Group | Standardized Implementation, Patients | Tailored Implementation, Patients | Standardized Implementation, Therapists | Tailored Condition, Therapists
Started | 39; 2 Health Clinics | 33; 2 Health Clinics | 28; 2 Health Clinics | 29; 2 Health Clinics
Completed | 26; 2 Health Clinics | 28; 2 Health Clinics | 28; 2 Health Clinics | 29; 2 Health Clinics
Not Completed | 13; 0 Health Clinics | 5; 0 Health Clinics | 0; 0 Health Clinics | 0; 0 Health Clinics
Not completed — Lost to Follow-up | 10 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0
Period: Clinics #11-12: Beginning Dec 2016
Arm/Group | Standardized Implementation, Patients | Tailored Implementation, Patients | Standardized Implementation, Therapists | Tailored Condition, Therapists
Started | 46; 1 Health Clinics | 19; 1 Health Clinics | 15; 1 Health Clinics | 23; 1 Health Clinics
Completed | 37; 1 Health Clinics | 17; 1 Health Clinics | 15; 1 Health Clinics | 23; 1 Health Clinics
Not Completed | 9; 0 Health Clinics | 2; 0 Health Clinics | 0; 0 Health Clinics | 0; 0 Health Clinics
Not completed — Lost to Follow-up | 6 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 12 clinics were assigned to standardized (n=6) or tailored (n=6) implementation. 228 patients (141 standardized, 87 tailored) are included in the analyses. Although patients and therapists were "assigned" to standardized or tailored implementation (depending on where they worked or received services), all analyses are at the participant-level (not site-level).
Groups:
- Standardized Implementation, Patients: Sites in this arm will receive the standard implementation of measurement based care intervention.
  Standard Implementation of Measurement Based Care: measurement based care in this study is the practice of basing psychotherapeutic services on the results of the Patient Health Questionnaire (PHQ-9), the implementation of measurement based care will be standardized such that clinicians will be encouraged to administer the PHQ-9 to depressed clients before each session.
- Tailored Implementation, Patients: Sites in this arm will receive the tailored implementation of measurement based care intervention.
  Tailored Implementation of Measurement Based Care: measurement based care in this study is the practice of basing psychotherapeutic services on the results of the Patient Health Questionnaire, the implementation of measurement based care will be tailored based on clinic specific barriers and facilitators.
- Standardized Implementation, Therapists: Sites randomized to the standardized condition will be expected to use the Patient Health Questionnaire prior to each session with a depressed client and they will work as a team to maximize fidelity.
- Tailored Implementation, Therapists: Sites randomized to the tailored condition will develop a site-specific protocol for use of the Patient Health Questionnaire and they will work as a team to maximize the fit of measurement based care to this clinic.
- Total: Total of all reporting groups
Arm/Group | Standardized Implementation, Patients | Tailored Implementation, Patients | Standardized Implementation, Therapists | Tailored Implementation, Therapists | Total
Number analyzed (Participants) | 141 | 87 | 71 | 83 | 382
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.06 (11.48) | 40.14 (11.74) | 45.23 (14.07) | 41.99 (13.22) | 41.32 (12.36)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Identity: Female | 96 | 61 | 54 | 67 | 278
  Gender Identity: Male | 44 | 26 | 17 | 15 | 102
  Gender Identity: Transgender | 0 | 0 | 0 | 1 | 1
  Gender Identity: Non-binary | 0 | 0 | 0 | 0 | 0
  Gender Identity: Missing | 1 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 15 | 3 | 0 | 31
  Not Hispanic or Latino | 127 | 70 | 67 | 83 | 347
  Unknown or Not Reported | 1 | 2 | 1 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 2 | 0 | 6
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 22 | 6 | 10 | 8 | 46
  White | 105 | 65 | 55 | 74 | 299
  More than one race | 2 | 1 | 2 | 1 | 6
  Unknown or Not Reported | 11 | 12 | 1 | 0 | 24
Region of Enrollment [Number; unit: participants]
  United States | 141 | 87 | 71 | 83 | 382
Highest Education Status [Count of Participants; unit: Participants]
  Some high school | 26 | 8 | 0 | 0 | 34
  High school diploma or equivalent | 54 | 30 | 0 | 0 | 84
  Some college, but no degree | 34 | 35 | 0 | 0 | 69
  Associate's degree | 9 | 5 | 0 | 0 | 14
  Bachelor's degree | 8 | 4 | 2 | 2 | 16
  Master's degree | 2 | 1 | 66 | 79 | 148
  Doctoral degree or equivalent | 2 | 0 | 2 | 1 | 5
  Other | 6 | 4 | 1 | 0 | 11
  Missing or not reported | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire
Description: Patient Health Questionnaire-9 (PHQ-9): screening tool for depression that can be used to monitor symptom change over time and inform care.
  Minimum value: 0 Maximum value: 27 Higher scores indicate a greater severity of depression (i.e., worse outcome).
Time Frame: Week 0 (baseline) and Week 12 of treatment
Population: In the standardized implementation condition, 141 patients provided baseline data and 102/141 participants provided 12-week data. In the tailored implementation condition, 87 patients provided baseline data and 74/87 provided 12-week data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Standardized Implementation: Sites randomized to the standardized condition will be expected to use the Patient Health Questionnaire prior to each session with a depressed client and they will work as a team to maximize fidelity. Sites in this arm will receive the standard implementation of measurement based care intervention.
  Standard Implementation of Measurement Based Care: measurement based care in this study is the practice of basing psychotherapeutic services on the results of the Patient Health Questionnaire (PHQ-9), the implementation of measurement based care will be standardized such that clinicians will be encouraged to administer the PHQ-9 to depressed clients before each session.
- Tailored Implementation: Sites randomized to the tailored condition will develop a site-specific protocol for use of the Patient Health Questionnaire and they will work as a team to maximize the fit of measurement based care to this clinic. Sites in this arm will receive the tailored implementation of measurement based care intervention.
  Tailored Implementation of Measurement Based Care: measurement based care in this study is the practice of basing psychotherapeutic services on the results of the Patient Health Questionnaire, the implementation of measurement based care will be tailored based on clinic specific barriers and facilitators.
Arm/Group | Standardized Implementation | Tailored Implementation
Number analyzed (Participants) | 141 | 87
score on a scale
  Baseline | 18.04 (4.10) | 16.77 (4.73)
  12-Week: number analyzed (Participants) | 102 | 74
  12-Week | 12.15 (6.07) | 13.09 (5.76)

2. Primary Outcome: PHQ-9 Completed Fidelity
Description: PHQ-9 fidelity was monitored for each individual psychotherapy session. Fidelity was scored as: (1) Therapist did not complete or record any PHQ-9 scores; (2) Therapist completed PHQ-9 and recorded scores in the EHR only; or (3) Therapist completed PHQ-9, recorded scores in the EHR, and discussed scores with the patient.
  The unit of measure is the number individual psychotherapy sessions conducted during the 5-month implementation window. Patient data were included for any patient at least 18 years old at the time of their first session with a participating therapist, regardless of if the patient was enrolled in the study.
Time Frame: 5-month implementation window
Population: For each participating therapist, the raw counts of fidelity (scored as 1, 2, or 3) are included at the session-level for the 15,686 individual psychotherapy sessions.
Measure: Count of Units; unit: Individual psychotherapy sessions
Units Other Than Participants: Individual psychotherapy sessions
Groups:
- Standardized Implementation, Therapists: Sites randomized to the standardized condition will be expected to use the Patient Health Questionnaire prior to each session with a depressed client and they will work as a team to maximize fidelity.
  Standard Implementation of Measurement Based Care: measurement based care in this study is the practice of basing psychotherapeutic services on the results of the Patient Health Questionnaire (PHQ-9), the implementation of measurement based care will be standardized such that clinicians will be encouraged to administer the PHQ-9 to depressed clients before each session
- Tailored Implementation, Therapists: Sites in the tailored condition arm will receive the tailored implementation of measurement based care intervention (PHQ-9).
  Tailored Implementation of Measurement Based Care: measurement based care in this study is the practice of basing psychotherapeutic services on the results of the Patient Health Questionnaire, the implementation of measurement based care will be tailored based on clinic specific barriers and facilitators
Arm/Group | Standardized Implementation, Therapists | Tailored Implementation, Therapists
Number analyzed (Participants) | 71 | 83
Number analyzed (Individual psychotherapy sessions) | 7570 | 8116
Individual psychotherapy sessions
  1. PHQ-9 Not Completed | 4894 | 5270
  2. PHQ-9 Completed (Reported in EHR) Only | 1564 | 860
  3. PHQ-9 Completed and Discussed with Patient | 1112 | 1986

ADVERSE EVENTS:
Time Frame: Collected during a client's enrollment in the study (i.e., approximately 12 weeks).
Description: Adverse events were only tracked and assessed for patients, not therapists. This was because, to the best of our knowledge, therapists were not likely to experience adverse events, as they were only making changes to their routine clinical practice. Patients, however, all had a depression diagnosis, were receiving clinical care, and were more sensitive to adverse events, such as medical hospitalization, suicidal ideation, or death.
Groups:
- Standardized Implementation, Patients: Sites randomized to the standardized condition will be expected to use the Patient Health Questionnaire prior to each session with a depressed client and they will work as a team to maximize fidelity. Sites in this arm will receive the standard implementation of measurement based care intervention.
  Standard Implementation of Measurement Based Care: measurement based care in this study is the practice of basing psychotherapeutic services on the results of the Patient Health Questionnaire (PHQ-9), the implementation of measurement based care will be standardized such that clinicians will be encouraged to administer the PHQ-9 to depressed clients before each session
- Tailored Implementation, Patients: Sites randomized to the tailored condition will develop a site-specific protocol for use of the Patient Health Questionnaire and they will work as a team to maximize the fit of measurement based care to this clinic. Sites in this arm will receive the tailored implementation of measurement based care intervention.
  Tailored Implementation of Measurement Based Care: measurement based care in this study is the practice of basing psychotherapeutic services on the results of the Patient Health Questionnaire, the implementation of measurement based care will be tailored based on clinic specific barriers and facilitators
Arm/Group | Standardized Implementation, Patients | Tailored Implementation, Patients
All-Cause Mortality (participants affected / at risk) | 0/141 | 1/87
Serious Adverse Events (participants affected / at risk) | 5/141 | 8/87
Other Adverse Events (participants affected / at risk) | 0/141 | 1/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standardized Implementation, Patients (N=141) | Tailored Implementation, Patients (N=87)
Suicidal Ideation (Psychiatric disorders) | 5 (5) | 7 (7)
Medical Hospitalization (Psychiatric disorders) | 0 (0) | 0 (0)
Death (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standardized Implementation, Patients (N=141) | Tailored Implementation, Patients (N=87)
Inappropriate Behavior Toward Staff (Psychiatric disorders) | 0 (0) | 1 (1) — e.g., threatening behavior/language

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT02266134/Prot_SAP_000.pdf
  • Informed Consent Form (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT02266134/ICF_001.pdf